CLINICAL TRIAL: NCT04526093
Title: MC-RWE : Real World Evidence in Patient-Reported Outcomes for Medical Cannabis: A Prospective Observational Study
Brief Title: Real-World Evidence in Patient-Reported Outcomes for Medical Cannabis (MC-RWE)
Acronym: MC-RWE
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Avicanna Inc (Industry)
Responsible Party: Principal Investigator, Jo Carroll, Research Manager, University Health Network, Toronto
Other Study IDs: 20-5537; 16560 (Other: Veritas IRB)
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pain; Sleep; Anxiety; Depression; Epilepsy
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression; Epilepsy | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical Cannabis — Verified medical cannabis products available within the current real-world study conform to Health Canada testing requirements
  Other Names: Medical Marijuana

SUMMARY:
This prospective observational study aims to describe the effectiveness of MC on pain, epilepsy, sleep and /or anxiety/depression in a cohorts of patients authorized to use MC, using pre-defined, validated self assessment scales.

DETAILED DESCRIPTION:
Given the recent legislative changes, medical cannabis has quickly garnered attention in clinical research as a potential pharmacotherapy to treat epilepsy, mood disorders, anxiety/depression disorders, sleep disorders and pain (neuropathic and non-cancer chronic pain)-conditions with often debilitating patient impact, substantive economic burden, and limited treatment options.

While there is growing evidence that MC may be an effective therapeutic option for patients suffering from chronic medical conditions, clinical research on medical cannabis has focused primarily on short-term outcomes, with limited attention to long-term benefits of specific strains, dosing regimens or treatment modalities. In addition, patients using MC generally are unable to maintain a defined treatment regimen (whether defined by strain name, biochemical composition, or mode of ingestion) over a long period of time. Even for patients desiring to maintain treatment with the same regimen, it may be impossible to do so, given the tendency for recreational and licensed medical producers to change their strains and product line up without notice. Such changes complicate MC users' efforts to optimize their overall health outcomes, as well as researchers' ability to study long-term effectiveness and safety of MC in general, and specific strains in particular.

Over the last few years, there has been an influx of new growers and an introduction of many new cannabis strains, each with a different representation of at least 500 known metabolites. Subtle changes in strain composition may have significant clinical effects. With so many strains available, and with limited information on strain composition and genetics, patients have little ability to control what they are taking over time.

The current real-world study addresses these complexities by providing patients verified MC strains and products, allowing them to maintain their treatment if desired or alter its composition in order to identify dosing regimens that work for them.

This study will provide much-needed pragmatic and objective information for patients and their clinicians about the effectiveness of verified MC products in the real-world setting using validated patient report outcome (PRO) tools.

The first study, of its kind in Canada, aims to recruit 1000 participants across the country. Digital patient consent will occur at the time of registration on the Avicanna's e-commerce platform(MyMedi.ca) when the study participant registers to purchase their MC and agrees to be part of the MC-RWE observational study.

Once a study participant is registered in the study and completed the baseline questionnaires, they will be given access to verified medical cannabis products (i.e., dried flower, oils, extracts and other cannabis product as they become approved and available) on the MyMedi.ca platform. Participants in the epilepsy group will be given access to verified medical cannabis products once they have completed baseline seizure frequency reporting at 6 weeks after enrollment in the study. This is a novel innovation within the Canadian Cannabis Industry.

Study participants will be administered a number of validated questionnaires upon study initiation, including an enrollment questionnaire that asks about medical history and specific questionnaires for pain, sleep, anxiety/depression. In addition, all participants will complete a health-related quality of life questionnaire.

All questionnaires will be self-administered online at time points Baseline, 6, 12, 18 (if applicable) and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (≥19 years of age) who are MC-naïve or -experienced with a medical authorization for MC provided by a prescribing health care practitioner and who have provided informed consent
* Primary therapeutic indications for MC use: pain, epilepsy, sleep, and/or anxiety/depression.
* Subjects agree to use verified products and refrain from using any other cannabis products, either medical or recreational, during the duration of the study

Exclusion Criteria:

* Concomitant use of illicit drugs
* Concomitant use of recreational cannabis

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Study participants (≥19 years of age) who are MC-naïve or -experienced with a medical document provided by a prescribing health care practitioner for the use of MC primarily for pain, epilepsy, sleep, and/or anxiety/depression.
  * Study participants who are either new or already registered with MyMedi.ca and consent to use verified products during the study.
  * Use of other cannabis products, either medical or recreational, is prohibited during the study period. Note: Although prohibited, the study cannot control for recreational cannabis use during the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to week 24 post-authorization of MC: Measured using the numerical rating scale (NRS). | Baseline, 6, 12, 18 (if applicable) and 24 weeks
  The 11-point NRS ranges from '0' being no pain to '10'' being the worst pain imaginable.
  Higher pain scores indicate greater pain intensity.
Change in pain interference from baseline to week 24 post-authorization of MC: Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS)-Pain Interference short form 6a. | Baseline, 6, 12, 18 (if applicable) and 24 weeks
  The PROMIS-short form 6a measures six items on 5-point scales (1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit and 5=very much) for pain interference on aspects of daily life. Scores are calculated from the total of item responses, with higher scores reflecting greater pain interference.
Sleep: Change in the Pittsburgh Sleep Quality Index (PSQI) from baseline to week 24 post-authorization of MC | Baseline, 6, 12, 18 (if applicable) and 24 weeks
  The PSQI contains 19-self rated questions and 5-questions rated by the roommate or bed partner. The 19 self-rated questions are combined to form seven component scores, each of which has a range of 0-3 points (0=no difficulty to 3=severe difficulty). Higher scores indicate worse sleep quality.
Anxiety: Change in the symptoms from baseline to week 24 post-authorization of MC; Measured using Generalized Anxiety Disorder 7-item scale (GAD-7). | Baseline, 6, 12, 18 (if applicable) and 24 weeks
  This 7-item scale assesses the signs of GAD (e.g. ''Feeling afraid as if something awful might happen") with response option of : 0= Not at all, 1=Several days, 2= More than half the days and 3= Nearly everyday. Scores are calculated from the total of item responses, with higher scores reflecting greater anxiety.
Depression: Change in the symptoms from baseline to week 24 post-authorization of MC. Measured by Patient Health Questionnaire 9 item scale (PHQ-9). | Baseline, 6, 12, 18 (if applicable) and 24 weeks
  The PHQ-9 assesses the signs of depression (e.g. Little interest or pleasure in doing things) with response option of : 0= Not at all, 1= Several days, 2= More than half the days, 3= Nearly everyday. Scores are calculated from the total of item responses, with higher scores reflecting the severity of depression.
Change in quality of life from baseline to Week 24: Measured using EuroQuol-5D-3-level health questionnaires(EQ-5D-3L) assessment scale. | Baseline, 6, 12, 18 (if applicable) and 24 weeks
  The EQ-5D-3L assesses health state in each of 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) on 3-point scale (no problems, some problems, extreme problems). Patients also rate their health on a vertical visual analogue scale with the endpoints "The best health you can imagine" and "The worse health you can imagine".
Epilepsy: change in seizure frequency for multiple different seizure types from baseline to Week 24 | Baseline, 6, 12, 18 and 24 weeks
  Seizure frequency will be documented in a patient diary, and number of seizures of each seizure type in the preceding 6 weeks will be reported.

SECONDARY OUTCOMES:
Demographics | Baseline
  Describe the demographic of patients (e.g. age, gender) authorized for MC in Canada using customized questionnaire.
Clinical characteristics of patients | Baseline
  Describe the Clinical characteristics (e.g. comorbidities, concomitant medications, etc.) of patients authorized for MC in Canada using customized questionnaire.
Patient satisfaction with the e-commerce platform's support team | 24 weeks after study initiation
  The qualitative value of using the e-commerce platform and support services to the overall patient experience, as assessed by a customized questionnaire
Changes in prescription medications of interest | 24 weeks after study initiation
  Change in use of concomitant medications (e.g., opioids, anti-depressants, anxiolytics, high-dosage anti-inflammatories, antiepileptic drugs) over time on study, assessed by customized questionnaire.

OTHER OUTCOMES:
The proportion of patients who have reported adverse effects due to MC use, as well as an assessment of the adverse effects based on different doses and methods of consumption. | 6,12, 18 (if applicable) and 24 weeks after study initiation
  A customized cannabis use questionnaire will be administered to collect information on side effects, dosage, and product types.
The proportion of patients who discontinued using MC during the course of the study as well the evaluation of the various reasons for this. | 6,12, 18 (if applicable) and 24 weeks after study initiation
  A customized cannabis use questionnaire will be administered to collect relevant information (i.e., when and why participants stopped using medical cannabis products, and if there is any leftover product, what they intended to do with it).

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD, PhD, Principal Investigator — Toronto General Hospital, UHN
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided